CLINICAL TRIAL: NCT05227963
Title: Comparison Between Soft Tissue Mobilization and Strengthening Exercises in Management of Local Neck Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Health Education Research Foundation (HERF) (Other)
Responsible Party: Principal Investigator, Javairia Javaid, Senior Physiotherapist, Health Education Research Foundation (HERF)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: Ref.No.Research/21
Record Dates: First submitted 2021-10-26; First posted 2022-02-08 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-01

CONDITIONS: Chronic Pain; Neck Pain
Keywords: Assessment; Neck pain; Pain measurements; Patient outcome assessment; Treatment outcome
MeSH Terms: conditions — Chronic Pain; Neck Pain

STUDY DESIGN:
Intervention Model Description: The randomized control study was conducted in two groups,one was experimental group received soft tissue mobilization and other was control group received strengthening exercises with supportive treatment for both groups.
Who Masked: Investigator
Masking Description: Non-probability convenient sampling technique was used to recruit the sample through lottery method into two groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group(Group A) (Experimental): Experimental Group received soft tissue mobilization with neck isometric strengthening exercises.
  Interventions: Other: soft tissue mobilization; Other: neck isometric strengthening exercises
- Control group (Group B) (Other): Control group received neck isometric strengthening exercises alone.
  Interventions: Other: neck isometric strengthening exercises

INTERVENTIONS:
Other: soft tissue mobilization — In this group, each participants received 45-minutes long session that includes 25-minutes of soft tissue mobilization and 20-minutes of neck isometric strengthening exercises. In each session, patient was seated on chair and sustained pressure, direct oscillation, perpendicular mobilization, parallel mobilization, and friction massage was applied on the neck musculature for a minute followed by a release for 30 seconds. This protocol was repeated three times in each session. Each session was repeated four-times a week for two-weeks (a total eight sessions).
  Arms: Experimental Group(Group A)
Other: neck isometric strengthening exercises — In this group, each participant received 20-minutes long session. Each session started in seated position and participants were asked to perform flexion, extension, side bending and rotation against resistance. During flexion movement, therapist placed hand on forehead and asked patient to move the neck forward, while in extension, therapist hand was placed at back of the head and patient had to move neck in backward direction. However, in side bending and rotation- therapist hand was placed at lateral side of the head and asked patient to side bend the neck and look at shoulder in the same direction respectively. Each session was repeated four-times a week for two-weeks (a total eight sessions).

SUMMARY:
A single-blinded, parallel-group randomized controlled trial was conducted at the national institute of rehabilitation medicine, Pakistan, from April to July 2016, on 30 females who were recruited through non-probability convenient sampling technique and randomly allocated to the experimental and control group.

DETAILED DESCRIPTION:
The experimental group received STM and neck isometric strengthening exercises, whereas the control group received neck isometrics strengthening exercises only. Numeric Pain Rating Scale (NPRS) was used to assess the pain intensity, while Neck Disability Index (NDI) was used to assess the neck-related disability. The data was collected pre-, during, and post-intervention. Repeated measure analysis of variance (RM ANOVA) was used to analyze within the group changes, while independent t-test was used to analyze the differences between the groups. Data were analyzed by using SPSS version 21.

This study describes the comparative effectiveness of STM when used as adjunct to strengthening exercises and when strengthening exercises are used alone for the management of TNS. According to the results of this study, STM in combination with neck isometric strengthening exercises as well as exercises alone were effective for managing neck pain and functional disability when a comparison was made within the groups.

ELIGIBILITY:
Inclusion Criteria

:• Age above 30 and below 75 years

* Patients having local neck pain included
* Female included
* With chronic neck syndrome (> month)

Exclusion Criteria:

* Age below 30 and more than 75 years
* Patients having radiating pain excluded
* Male excluded.
* With acute neck syndrome (< 3 month)

Ages: 30 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-04-04 (Actual); Primary Completion 2016-05-10 (Actual); Study Completion 2021-08-20 (Actual)

PRIMARY OUTCOMES:
Numerical pain rating scale (NPRS) | upto 2 weeks
  NPRS was used to assess the pain intensity. The 11-point numeric scale ranging from 0-10; 0 means no pain while 10 means worst possible pain.
Neck disability index (NDI) | upto 2 weeks.
  NDI was used to assess the neck-related disability. Of the 50 score, 0-4 means no disability while 35-50 means severe disability.
Neck range of motion | upto 2 weeks .
  Goniometer was used to measure the range of motion of neck.

IPD SHARING:
Plan to Share IPD: No